CLINICAL TRIAL: NCT07164547
Title: Acute Effects of Tribulus Terrestris Supplementation on Anaerobic Performance and Sprint Times in Combat Sport Athletes: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial
Brief Title: Acute Effects of Tribulus Terrestris on Anaerobic Power and Sprint Performance in Combat Sport Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salih ÇABUK (Other)
Responsible Party: Sponsor-Investigator, Salih ÇABUK, Research Assistant, Erzurum Technical University
Organization: Erzurum Technical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETU-TRIBULUS-2025; E-70400699-050.02.04-250010269 (Other: Ataturk University)
Record Dates: First submitted 2025-08-31; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Anaerobic Power; Sprint Performance
Keywords: Tribulus terrestris; Combat sports; Anaerobic performance; Wingate test; Sprint time; Ergogenic supplementation
MeSH Terms: interventions — Tribulus extract; Cellulose

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, crossover trial in which all participants received both Tribulus terrestris and placebo supplementation with a wash-out period in between conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, care providers, and outcome assessors were blinded to group allocation. Supplements were prepared in identical capsules to ensure blinding integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tribulus Terrestris (Experimental): A single oral dose of 625 mg Tribulus terrestris extract (40% saponins) given 60 minutes before exercise testing.
  Interventions: Dietary Supplement: Tribulus terrestris extract
- Placebo (Placebo Comparator): Visually identical cellulose capsule given 60 minutes before exercise testing.
  Interventions: Other: Cellulose capsule (placebo)

INTERVENTIONS:
Dietary Supplement: Tribulus terrestris extract — 625 mg oral capsule (40% saponins), single dose
  Arms: Tribulus Terrestris
Other: Cellulose capsule (placebo) — Oral cellulose capsule, identical in appearance
  Arms: Placebo

SUMMARY:
This study aims to investigate the acute effects of Tribulus terrestris supplementation on anaerobic performance and sprint times in trained male combat sport athletes. A total of 28 athletes from kickboxing, Muay Thai, and taekwondo disciplines will participate in a randomized, double-blind, placebo-controlled, crossover trial.

Participants will ingest either a single oral dose of 625 mg Tribulus terrestris (40% saponins) or a placebo 60 minutes before performing performance tests. The performance assessments will include a 30-second Wingate anaerobic cycling test and 20 m and 100 m sprint tests using photocell timing gates. After a wash-out period, participants will cross over to the alternate condition.

The primary outcomes are peak power and mean power from the Wingate test and sprint times over 20 m and 100 m.

DETAILED DESCRIPTION:
This trial is designed to evaluate the acute ergogenic potential of Tribulus terrestris supplementation in combat sport athletes. Tribulus terrestris has traditionally been marketed as a natural testosterone booster and performance enhancer, yet its acute effects on high-intensity exercise performance remain unclear.

Design and Methods

Participants: 28 trained male athletes (Kickboxing n=12, Muay Thai n=10, Taekwondo n=6), aged 18-30 years, with at least 2 years of competitive training experience.

Design: Randomized, double-blind, placebo-controlled, crossover.

Intervention: A single dose of 625 mg Tribulus terrestris (40% saponins) or matched placebo (cellulose). Supplements will be ingested 60 minutes before testing.

Procedures: After a standardized warm-up, participants will complete a 30-second Wingate test on a Monark cycle ergometer (resistance = 10% body mass) to measure peak power, mean power, and fatigue index. Following 10 minutes of recovery, participants will perform 20 m and 100 m sprint tests using double-beam photocells (Witty timing system). Each participant will perform both supplementation conditions with a ≥72 h wash-out.

Outcomes Primary outcomes: Wingate peak power (W, W/kg), mean power (W, W/kg). Secondary outcomes: 20 m and 100 m sprint times (s).

Ethics: Approved by the Ethics Committee of Atatürk University (Protocol No: E-70400699-000-2500104927). Written informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged 18-30 years
* Engaged in combat sports (kickboxing, Muay Thai, or taekwondo)
* Minimum 2 years of continuous training experience
* Training at least 4 sessions per week
* Free from injury or illness at the time of testing
* Provided written informed consent

Exclusion Criteria:

* Use of ergogenic supplements, anabolic steroids, or hormonal treatments within the past 3 months
* Consumption of caffeine, alcohol, or performance-enhancing substances within 24 hours before testing
* Current musculoskeletal injury or medical condition that may limit performance
* Any chronic disease or contraindication to high-intensity exercise

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Peak Power Output (W, W/kg) - Wingate Test | Measured once, 60 minutes after supplementation, during the Wingate test session (single-day assessment).
  Maximum anaerobic power generated during the 30-second Wingate cycling test performed against a resistance equal to 10% of body mass.

SECONDARY OUTCOMES:
Mean Power Output (W, W/kg) - Wingate Test | Measured once, 60 minutes after supplementation, during the Wingate test session (single-day assessment).
  verage anaerobic power calculated across the full 30-second Wingate cycling test.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Sports Science Laboratory, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Plan Description: If shared, the de-identified individual participant data (IPD) will include Wingate anaerobic test outcomes and sprint performance times. These data represent the analyzable dataset collected during the study. If data are not shared, this will be due to limitations related to participant confidentiality and data protection.
  Access Criteria: Data may be made available upon reasonable request from qualified researchers for academic, non-commercial purposes. Requests will be reviewed by the study investigators, and data will only be shared after publication of the primary results.